CLINICAL TRIAL: NCT02249143
Title: Duration of Continuous Positive Airway Pressure and Pulmonary Function Testing in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cynthia McEvoy, Professor of Pediatrics, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eIRB00010607
Record Dates: First submitted 2014-08-28; First posted 2014-09-25 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: Continuous positive airway pressure; Prematurity; Respiratory distress syndrome; Bronchopulmonary dysplasia
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Premature Birth | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP and room air (Active Comparator): Stable premature infants on CPAP and room air will be randomized to stay on CPAP for an additional two weeks.
  Interventions: Device: CPAP and room air
- Room air (No Intervention): Premature stable infants on CPAP and room air will be randomized to transition to room air alone.

INTERVENTIONS:
Device: CPAP and room air — Stable premature infants on CPAP and room air and meeting specific stability criteria will be randomized to stay on continuous positive airway pressure and room air for an additional two weeks or will be transitioned to room air alone.
  Other Names: continuous positive airway pressure
  Arms: CPAP and room air

SUMMARY:
The primary aim of this study is to quantify and compare changes in lung volumes (as measured by functional residual capacity) in premature infants stable on continuous positive airway pressure (CPAP), and then randomized to two additional weeks of CPAP and room air versus room air alone. We hypothesize that infants randomized to additional CPAP will demonstrate an increased functional residual capacity (at the end of the two week study period and prior to discharge) compared to those randomized to room air.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth <33 weeks
* Required CPAP for a minimum of 24 hours for respiratory distress
* Patient on CPAP and room air at time of randomization

Exclusion Criteria:

* Complex congenital heart disease other than patent ductus arteriosus or atrial septal defect
* Major malformations or chromosomal anomalies
* Multiple gestation greater than twins
* Culture proven sepsis or unstable at time of randomization

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy T McEvoy, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Lam R, Schilling D, Scottoline B, Platteau A, Niederhausen M, Lund KC, Schelonka RL, MacDonald KD, McEvoy CT. The Effect of Extended Continuous Positive Airway Pressure on Changes in Lung Volumes in Stable Premature Infants: A Randomized Controlled Trial. J Pediatr. 2020 Feb;217:66-72.e1. doi: 10.1016/j.jpeds.2019.07.074. Epub 2019 Sep 10. PMID 31519441

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPAP and Room Air | Room Air
Started (randomized) | 24 | 26 (randomized)
Completed | 22 (with technically acceptable pulmonary function tests in the neonatal intensive care unit) | 22 (with technically acceptable pulmonary function tests in the neonatal intensive care unit)
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: CPAP and Room Air: CPAP and room air: Stable premature infants on CPAP and room air and meeting specific stability criteria will be randomized to stay on continuous positive airway pressure and room air for an additional two weeks or will be transitioned to room air alone.
- No Intervention: Room Air: Premature stable infants on CPAP and room air will be randomized to transition to room air alone.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: CPAP and Room Air | No Intervention: Room Air | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 9 | 14 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Measurements of Functional Residual Capacity (FRC) in Randomized Premature Infants
Description: Functional residual capacity (FRC) was measured with the nitrogen washout technique. For the nitrogen washout technique, calibration is done with 2 known volumes, and a calibration line was constructed for the system at the specific flow rate and used to correlate the nitrogen washed out to the infant's FRC. The system corrected for dead space and corrected the FRC to body temperature, pressure, and water-saturated conditions. Acceptance criteria included: 1) infant supine and quietly asleep; 2) test initiated at end expiration; 3) no evidence of leak on tracing of the washout; 4) consistent tracings; 5) at least 2-3 measurements with a coefficient of variation <10%. These are testing and acceptance criteria outlined by the American Thoracic Society and European Respiratory Society.
Time Frame: Just prior to randomization, two weeks later and at discharge (an average of 34 to 37 weeks of corrected gestational age).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
mL
  FRC change from baseline to two weeks | 12.6 (11.4) | 6.4 (10.1)
  FRC change from baseline to discharge | 27.2 (12.5) | 17.1 (11.7)
Statistical Analysis 1: Comparison: CPAP and Room Air vs Room Air; FRC values over time were modeled using linear mixed effects regression with treatment group vs. time interaction and repeated measures for the randomization, 2 week, and discharge time points. Compound symmetric covariance structures were used to account for the correlation of FRC values within each patient. We compared outcomes between the two treatment groups and included adjustments for gender, twin gestation, and weight at randomization; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Net) = 6.62, 95% CI 2-sided [0.02 to 13.22]

2. Secondary Outcome: Measurements of Passive Respiratory Compliance in Randomized Premature Infants
Description: Measurements of passive respiratory compliance will be done with the single breath occlusion technique.
Time Frame: Just before randomization, two weeks later, and at discharge at about 35-37 weeks of corrected gestational age
Measure: Mean (Standard Deviation); unit: mL/Kg
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
mL/Kg
  At Randomization | 1.37 (0.28) | 1.32 (0.28)
  At End of 2 Weeks of Treatment | 1.28 (0.28) | 1.17 (0.18)
  At Discharge | 1.08 (0.18) | 1.12 (0.21)
Statistical Analysis 1: Comparison: CPAP and Room Air vs Room Air; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: CPAP and Room Air vs Room Air; Group differences in the secondary outcomes were tested at randomization, two weeks, and discharge using independent samples t-tests; Test type: Superiority

3. Secondary Outcome: Passive Respiratory Resistance in Randomized Premature Infants
Description: Measurements of passive respiratory resistance will be done with the single breath occlusion technique.
Time Frame: Just prior to randomization, two weeks after randomization, and at discharge at about 35-37 weeks of corrected gestational age.
Measure: Mean (Standard Deviation); unit: cmH2O/mL/sec
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
cmH2O/mL/sec
  At Randomization | 0.054 (0.014) | 0.053 (0.009)
  At End of 2 Weeks of Treatment | 0.061 (0.014) | 0.074 (0.021)
  At Discharge | 0.073 (0.02) | 0.082 (0.022)

4. Secondary Outcome: Measurements of Tidal Flow Volume Loops Will be Done in the Randomized Premature Infants.
Description: Characteristics of tidal flow volume loops will be measured.
Time Frame: Just before randomization, two weeks later, and at discharge at about 35-37 weeks of corrected gestational age.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
mL
  At Randomization | 7.1 (1.1) | 7.8 (0.97)
  At End of 2 Weeks of Treatment | 7.6 (1.1) | 7.4 (0.9)
  At Discharge | 7.3 (1.1) | 7.3 (0.56)

5. Other Pre Specified Outcome: Changes in the Growth Parameters Between the Randomized Premature Infants
Description: Changes in growth parameters will be compared between randomized groups.
Time Frame: From randomization through discharge at about 35-37 weeks of corrected gestational age.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
g
  At Randomization | 1567 (293) | 1482 (323)
  At Discharge | 2282 (354) | 2253 (413)

6. Other Pre Specified Outcome: The Number of Participants With Adverse Events and Serious Adverse Events in the Randomized Groups of Premature Infants.
Description: Adverse events and serious adverse events occurring in the randomized groups will be documented carefully
Time Frame: From randomization through discharge from the neonatal intensive care unit (an average of 35 to 37 weeks of corrected gestational age).
Measure: Number; unit: participants
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
participants | 0 | 0

7. Other Pre Specified Outcome: Corrected Gestational Age at Which Full Nipple Feeds Are Achieved
Description: The corrected gestational age at which full nipple feeds are achieved will be compared between the randomized groups.
Time Frame: Randomization through discharge at about 35-37 weeks of corrected gestational age.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
weeks | 35.9 [35.1 to 37.5] | 35.5 [34.7 to 37.0]

8. Other Pre Specified Outcome: Incidence of Wheezing Through One Year of Age
Description: Incidence of wheezing will be compared through one year of corrected gestational age between the randomized groups.
Time Frame: Discharge through one year of corrected age
Population: Number of participants analyzed is lower here as we were not able to follow all infants through 1 year of corrected age.
Measure: Count of Participants; unit: Participants
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 18 | 21
Participants | 7 | 6

9. Other Pre Specified Outcome: Cost Comparison Between Randomized Groups
Description: Cost comparison through 12 months of corrected gestational age between the randomized groups per percent improvement in FRC measured at discharge between the groups.
Time Frame: Through 12 months of corrected age
Population: Data not collected
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Days on Oxygen Between the Randomized Groups
Description: The days of oxygen supplementation will be compared between the groups of randomized patients.
Time Frame: Through discharge at about 35-37 weeks of corrected gestational age
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 22 | 22
days | 0 [0 to 2.3] | 0 [0 to 4.5]

11. Other Pre Specified Outcome: Days in the Hospital
Description: The days in the hospital will be compared between the randomized groups.
Time Frame: Delivery through discharge at about 35-37 weeks of corrected gestational age
Population: Data not collected
Arm/Group | CPAP and Room Air | Room Air
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CPAP and Room Air | Room Air
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No